CLINICAL TRIAL: NCT02591277
Title: A Prospective Observational Post-Marketing Study of Harvoni in Japanese Patients With Genotype 1 Chronic Hepatitis C Infection
Brief Title: Use-Results Surveillance Study of Harvoni® in Japanese Patients With Chronic Genotype 1 Hepatitis C Virus Infection
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-337-1498
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus; observational; post-marketing; ledipasvir/sofosbuvir; Japan
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Harvoni: Adult patients with chronic genotype 1 HCV infection with or without compensated cirrhosis who take Harvoni as part of routine clinical care at a participating clinic/hospital.
  Interventions: Drug: Harvoni

INTERVENTIONS:
Drug: Harvoni — Harvoni (90/400 mg) FDC tablet administered orally once daily
  Other Names: LDV/SOF; GS-5885/GS-7977

SUMMARY:
This study will evaluate the safety and efficacy of Harvoni® (ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC)) treatment under real world use in Japan. Among adult patients with chronic genotype 1 hepatitis C virus (HCV) infection and treated with Harvoni in routine clinical use, the primary objective of this study is to evaluate the incidence of adverse drug reactions (ADRs) under real world settings.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult patients with chronic genotype 1 HCV infection with or without compensated cirrhosis
* Patients who are prescribed Harvoni

Key Exclusion Criteria:

* None

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic genotype 1 HCV infection with or without compensated cirrhosis who take Harvoni as part of routine clinical care at a participating clinic/hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3294 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reaction (ADR) under real world settings | Up to 16 weeks

SECONDARY OUTCOMES:
Proportion of participants with sustained virologic response (SVR) 12 and 24 weeks after discontinuation of therapy (SVR12 and SVR24) | Posttreatment Weeks 12 and 24
  SVR12 and SVR24 are defined as HCV RNA < the lower limit of quantification (LLOQ) 12 and 24 weeks following the last dose of study drug, respectively.
Proportion of participants with HCV NS5A and NS5B resistance associated variants among patients who do not achieve SVR at 12 weeks | Approximately 12 weeks after treatment completion or discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (125):
- Japan (125):
  - Ageo-shi
  - Akita
  - Amagasaki-shi
  - Aomori
  - Arao-shi
  - Asahi-shi
  - Asahikawa-shi
  - Asakura-shi
  - Bunkyō City
  - Chiba
  - Chichibu-shi
  - Chuo-shi
  - Fujioka-shi
  - Fukui-shi
  - Fukuoka
  - Gifu
  - Hakodate-shi
  - Hamamatsu
  - Handa-shi
  - Hashima-shi
  - Hatsukaichi-shi
  - Higashiibaraki-gun
  - Hirosaki-shi
  - Hiroshima
  - Hitachi-shi
  - Hukui-shi
  - Ichikawa-shi
  - Iizuka-shi
  - Ikeda-shi
  - Inashiki-gun
  - Inzai-shi
  - Iruma-gun
  - Ise-shi
  - Iwaki
  - Izumo-shi
  - Izunokuni-shi
  - Kagoshima
  - Kamogawa-shi
  - Kanazawa
  - Karatsu-shi
  - Kashihara-shi
  - Kashiwa-shi
  - Kasukabe-shi
  - Kawagoe-shi
  - Kawaguchi-shi
  - Kawasaki-shi
  - Kirishima-shi
  - Kitakyushu-shi
  - Kitamoto-shi
  - Kobe
  - Kodaira-shi
  - Kofu
  - Komae-shi
  - Komaki-shi
  - Koriyama-shi
  - Koshigaya-shi
  - Kōtoku
  - Kuga-gun
  - Kuki-shi
  - Kumamoto
  - Kurashiki-shi
  - Kure-shi
  - Kurume-shi
  - Kyoto
  - Maebashi
  - Matsumoto-shi
  - Matsuyama
  - Minatoku
  - Miyazaki
  - Moriguchi-shi
  - Morioka
  - Nagakute-shi
  - Nagasaki
  - Nagoya
  - Nakagami-gun
  - Nerima-ku
  - Niigata
  - Nishinomiya-shi
  - Noshiro
  - Obihiro-shi
  - Ofukeshi
  - Okayama
  - Osaka
  - Osakasayama-shi
  - Oume-shi
  - Ōita
  - Ōmihachiman
  - Ōta-ku
  - Ōtsu
  - Saga
  - Saitama-shi
  - Sakaishi
  - Sano-shi
  - Sapporo
  - Sasebo-Shi
  - Sendai
  - Shimonoseki-shi
  - Shimotsuga-gun
  - Shimotsuke-shi
  - Shinagawa-ku
  - Shinjuku-ku
  - Shirakawa-shi
  - Shizuoka
  - Shunan-shi
  - Sumida-ku
  - Tagawa-shi
  - Takamatsu
  - Takasaki-shi
  - Toda-shi
  - Tokorozawa-shi
  - Tokushima
  - Tonami-shi
  - Toyama
  - Toyoake-shi
  - Ureshino-shi
  - Utsunomiya
  - Wakayama
  - Yachiyo-shi
  - Yamagata
  - Yanagawa-shi
  - Yatsushiro-shi
  - Yokkaichi-shi
  - Yokohama
  - Yonago-shi
  - Yoshida-gun

REFERENCES:
- [Derived] Mizokami M, Liu LJ, Fujiyama N, Littman M, Yuan J, Sekiya T, Hedskog C, Ng LJ. Real-world safety and effectiveness of ledipasvir/sofosbuvir for the treatment of chronic hepatitis C virus genotype 1 in Japan. J Viral Hepat. 2021 Jan;28(1):129-141. doi: 10.1111/jvh.13395. Epub 2020 Sep 16. PMID 32869924